CLINICAL TRIAL: NCT03080584
Title: Effect of 12 Weeks of Acupuncture on AMH and Ovarian Reserve in Women With Low Ovarian Reserve. A Pilot Study
Brief Title: Effect of 12 Weeks of Acupuncture on AMH and COH in Low Responder Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dansk Fertilitetsklinik (Other)
Responsible Party: Principal Investigator, Ursula Bentin-Ley, Physician, Dansk Fertilitetsklinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-16033980
Record Dates: First submitted 2017-02-28; First posted 2017-03-15 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Hypogonadism; Ovarian; Female Infertility
Keywords: acupuncture; IVF; AMH; ovarian reserve
MeSH Terms: conditions — Hypogonadism; Infertility, Female | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: comparison of AMH and ovarian response before and after acupuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acupucture arm (Experimental): all participants undergo 12 weeks of acupuncture
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — 12 weeks of acupuncture comprising basic acupuncture, ear acupuncture and Moving cups. On top of the basic acupuncture, additional locations can be added.

SUMMARY:
the investigators want to study whether 12 weeks of acupuncture has any effect on AMH and the ovarian reserve in women with low ovarian reserve (low responders). AMH is measured before and after 12 weeks of acupuncture and the clinical response to controlled ovarian hyperstimulation before and after the acupuncture is compared.

DETAILED DESCRIPTION:
AMH is measured cycle day 2 or 3 before and after 12 weeks of acupuncture and the levels are compared. Furthermore, secondary outcomes from IVF treatments before and after the intervention are compared.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ICSI treatment
* 18-40 years
* AMH measured < or = 10 pmol/l
* maximum of 8 oocytes collected at last treatment before inclusion-

Exclusion Criteria:

* (use of testicular sperm)
* more than 4 acupuncture treatments within the last 3 months before inclusion -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11-12 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
AMH | chance from baseline after 12 weeks of acupuncture
  anti-Müllerian Hormone level

SECONDARY OUTCOMES:
No. of oocytes aspirated | change from baseline treatment and after 12 weeks of acupunture
  the number of oocytes collected during egg aspiration for IVF
FSH dose/oocyte collected | change from baseline treatment and after 12 weeks of acupuncture
TQE 44 hours after fertilisation | change from baseline treatment and after 12 weeks of acupuncture
  The number of top quality embryos 44 hours after fertilisation
biobank with blood plasma | 2 years after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Bentin-Ley, M.D., Principal Investigator — Dansk Fertilitetsklinik
Locations (1):
- Dansk Fertilitetsklinik, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No